CLINICAL TRIAL: NCT00204594
Title: Local Treatment of Metastatic Melanoma With Autologous Lymphocytes and the Bispecific Antibody rM28
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Thomas Eigentler, Study Coordinator, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rM28-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Malignant Melanoma
Keywords: mRNA; vaccination; melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibody (Experimental)
  Interventions: Drug: rM28; Drug: autologous PBMCs

INTERVENTIONS:
Drug: rM28
Drug: autologous PBMCs

SUMMARY:
Phase I/II clinical trial to analyze safety and efficiency of intralesional application of the bispecific single chain antibody rM28 and autologous PBMCs in patients with metastatic melanoma stage III/IV and unresectable metastasis.

DETAILED DESCRIPTION:
Phase I/II clinical trial to analyze safety and efficiency of intralesional application of the bispecific single chain antibody rM28 and autologous PBMCs in patients with metastatic melanoma stage III/IV and unresectable metastasis. The antibody is directed against epitops of human CD28 and the melanoma associated surface antigen HMV-MAA. Treatment over 5 days with dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* malignant melanoma stage III/IV
* injectable soft tissue metastasis
* informed consent given
* Karnofsky >= 70%

Exclusion Criteria:

* additional chemotherapeutical treatment
* systemic glucocorticoids
* brain metestasis
* other malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
toxicity
clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Garbe Claus, Prof. Dr., Principal Investigator — Department of dermatology, university of tuebingen; Gundram Jung, Prof. Dr., Principal Investigator — University of Tuebingen, Dept. of Immunology
Locations (1):
- University of Tuebingen, Department of dermatology, Tübingen, Germany